CLINICAL TRIAL: NCT06443190
Title: Wichitasowin: Indigenous Patient Navigator for Young Adults Study
Acronym: Wichitasowin
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00138085
Record Dates: First submitted 2024-05-23; First posted 2024-06-05 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Chronic Diseases in Adolescence
Keywords: transition; Indigenous; community based participatory action research; health care navigator

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Indigenous Patient Navigator Support (Experimental): Participants will work with an Indigenous Patient Navigator (IPN) for up to 18 months. The IPN may have the following roles in supporting the youth +/- their caregiver in managing their healthcare and health condition:
  * Spiritual: connect with community Elders, connect with cultural programs, arrange smudging and ceremony
  * Physical: find housing, find a family doctor, arrange transportation, fill prescriptions, create a health passport
  * Mental: arrange health benefits, schedule appointments, find employment, connect to community services
  * Emotional: connect with peers, find mental health supports, support youth at appointments, communicate with youth's healthcare team
  Interventions: Other: Indigenous Patient Navigator Support

INTERVENTIONS:
Other: Indigenous Patient Navigator Support — See Arm Description

SUMMARY:
The objective of this pathway is to establish and evaluate a novel Indigenous-led patient navigator (IPN) program for Indigenous adolescents living with chronic health conditions in Maskwacis, Alberta. Over the last three years a community-based participatory research partnership was developed with Elders and community members from Maskwacis, Maskwacis Health Services, and researchers from the University of Alberta. Previous research identified the need for an IPN to support Indigenous young adults and their caregivers in managing their health conditions transitioning into adulthood and transferring from pediatric to adult healthcare. The aim of partnership now is to evaluate whether a community-derived IPN program co-designed with an established group of Maskwacis Elders, Knowledge Keepers, healthcare providers, caregivers and youth with lived experience can aid in improving the experience of transitioning into adult healthcare services for Indigenous youth and their families living in Maskwacis, Alberta.

DETAILED DESCRIPTION:
Purpose: to implement and evaluate a novel Indigenous Patient Navigator (IPN) pathway for Indigenous young adults with complex and chronic medical conditions, and their families, living in Maskwacis, AB learning to manage their health condition transitioning into adulthood.

Hypothesis: the Indigenous-Led Pathway for Young Adults will provide substantial benefits to youth and families, including but not limited to cultural ceremony and Elder-support, emotional support, accessing medical appointments and preventing loss to follow-up, feeling engaged with the adult health care system, developing self-management and self-advocacy skills, and reducing feelings of anxiety and isolation. The investigators expect the pathway will improve the health of Indigenous adolescents and young adults living with chronic health conditions in Maskwacîs, ultimately improving the wellbeing of the entire community.

Justification: The investigators' previous research has identified key barriers to care included finances (e.g., cost and availability of transportation to healthcare appointments), intergenerational trauma making it difficult to prioritize the health condition, racism and discrimination in health care settings, lack of cultural safety, and loss of benefits at age 18 (e.g., Jordan's Principle does not apply to young adults). Facilitating factors identified include family support and culture, peer support networks, health condition education, and having safe spaces in healthcare settings where Indigenous imagery and medicines were visibly displayed.

During a series of in-person meetings with our Community Advisory Committee (CAC) the Investigators discussed study findings and possible strategies to address them. The Elders and Knowledge Keepers concluded that a community-based, Indigenous-led patient navigator service would be a logical approach to helping transition-age youth navigate the healthcare system between pediatric and adult care. It was felt that both the barriers and facilitators summarized above provided evidence for the need for an IPN, and that an IPN could help mitigate some of the social determinants of health that prevent adolescents and young adults from attending medical appointments, filling prescriptions, and managing their health condition(s). IPN programs in Canada exist in acute care settings, children's hospitals, cancer care, and adult outpatient settings. To the Investigators' knowledge, a community based IPN program focusing on transition age youth does not yet exist in Canada.

Objectives

1. To strengthen the existing partnership with the CAC and Maskwacis Health Services, through regular gatherings, engaging in ceremony and traditions, respecting cultural protocol, encouraging feedback, and ensuring our committee members guide the project's activities to benefit the community in a good way.
2. To co-design and implement a novel IPN service for Indigenous adolescents with special health care needs residing in Maskwacis through community engagement sessions and meetings with senior management of Maskwacis Health Services and Alberta Health Services.
3. To evaluate the IPN service, addressing the following questions:

   1. How do Indigenous youth transitioning into adult care describe their experiences of transitioning, the role of the IPN in helping them through this transition, and the impact of the IPN program on the Indigenous perspective of health and wellness?
   2. How can these findings promote improved outcomes for Indigenous youth in transition?
4. To create sustainability of the IPN role within the Maskwacis community and enable the creation of an IPN program for transition-age youth in other Indigenous communities in Alberta, both on- and off-reserve.

Research Method/Procedures

Study design and setting: Qualitative study to evaluate an IPN program using a community-based participatory action research approach. The study will be conducted with and within the community of Maskwacis, Alberta, Maskwacis Health Services and the Awasisak Indigenous Health Program at the Stollery Children's Hospital. Maskwacis is located approximately 90 km southeast of Edmonton. It has a population of ~18 000 residents divided among Four Nations (Samson, Louis Bull, Ermineskin, Montana) and a small satellite location in Pigeon Lake.

Participant Recruitment: The CAC and community members will assist Investigators to find ways to recruit participants from the community. A community-based research assistant (RA) will approach potentially eligible participants at participating recruitment clinics.

IPN Role: The IPN role will be co-designed and implemented based on thorough community engagement including the CAC, Alberta Health Services and Maskwacis Health Services. Allowing flexibility within the role and developing the IPN role with guidance from the CAC and community will allow the IPN to serve participants, families and the community in the most appropriate and effective way.

Below is a list of supports that may potentially be provided to participants by the IPN:

1. Connect participants with community supports including housing, social assistance, disability payments, education, and employment opportunities.
2. Connect participants with cultural resources: cultural programming and events, ceremony, connection with Elders.
3. Scheduling primary care and/or specialty care appointments as appropriate to address specific medical/mental health needs.
4. Accessing transportation to medical and social service appointments.
5. Providing in person support and advocacy for participants during health care appointments.
6. Work with the participant to create a smart phone-based health passport containing key information about their health condition, names and doses of medications, schedule of upcoming appointments, and contact names, phone number and addresses for their doctors, nurses, and allied health professionals. For participants not having access to a smartphone, this information will be provided on a wallet-sized card.
7. Support adherence to follow-up clinic visits and health maintenance including completing clinically indicated laboratory tests and obtaining prescription refills as needed.
8. Assist with financial and insurance paperwork (e.g., Jordan's Principal, Non-Insured Health Benefits, Alberta Income for the Severely Handicapped).
9. Promote self-management skills by providing tools, educational resources, and coaching.
10. Facilitate in-person group sessions open to all participants at a community hall. Group sessions reduce isolation, empower youth to build connections, advocate for themselves and each other, and incorporate Indigenous cultural ceremonies.

Navigators will use electronic technology (cell phone, email, text message, social media) to maintain contact and provide support for participants. The needs of each participant will vary and hence the program will be participant and family-centered and specific. There will be no a priori limits on the frequency of contact between the navigator and participant; contact may be as frequent as daily, or as infrequently as every 2 months at a minimum, depending on participants' needs.

Health Information Access + Documentation:

Participants will be asked for permission for the research team and IPN to review their health information within their Electronic Medical Record within Alberta Health Services and Maskwacis Health Services databases, so the IPN can understand their health condition and how they use the health care system during this transition. The IPN will record every contact and nature of assistance provided using the AHS EMR Connect Care, in a standardized encounter format.

IPN training: Plan for an Indigenous identifying individual who has a minimum of a Bachelor of Social Work or a Bachelor of Science in Nursing, and experience working with adolescents and/or young adults in a community setting. The IPN will be trained by a) other IPNs in Alberta (e.g., Four Winds Program, led by team member Dr. Oster), b) staff at the Awasisak Indigenous Health Program at the Stollery with AHS onboarding and orientation as appropriately determined by the reporting manager, c) a non-Indigenous patient navigator at the Stollery, affiliated with the Transition Navigator Trial led by team member Dr. Mackie, and d) staff at Maskwacis Health Services. The IPN will receive privacy and confidentiality training as per TCPS-2, as well as AHS Privacy and Confidentiality Training. Most importantly, the IPN will be continually involved with the team's CAC to receive guidance and feedback on the IPN role and implementation and engage in ceremony.

Study Logistics:

1. Navigator Meeting: The IPN will schedule a face-to-face meeting with the participant, or with caregiver(s) if the participant has developmental delay precluding their participation independent of a caregiver, or both. Prior to the meeting the IPN will review the electronic medical record of the youth participant to understand their health condition and access of healthcare. During this meeting the IPN will complete an assessment of the participant's healthcare needs and learn about the participant's journey with their health condition, as well as build trust and rapport with the family. Using the information from both the interview, as well as from review of their electronic medical record, the navigator will create an individual-centered transition plan, in collaboration with the participant, caregiver(s), and if needed with community partners.
2. Navigator support: Participants will then work with the IPN for up to 18 months. Support offered by the IPN is previously described under "IPN Role".
3. Peer Support Sessions + Talking Circles: The IPN will organize peer support sessions for study participants held every 3 months in-person in Maskwacis. Both youth participants and caregiver participants are invited to take part in peer support sessions. The purpose of these sessions will be to build a sense of community for youth living with chronic health conditions and their caregivers, reduce isolation, and empower participants to develop self-management and self-advocacy skills together in an engaging and fun environment. Life skills topics such as budgeting and job interviewing will be included. A community Elder will attend the peer sessions to provide cultural ceremony and share traditional teachings such as smudging and prayer. During the sessions talking circles will be offered for participants to engage in discussion with Elders and each other regarding their experience working with the IPN. Participants may attend as many or as little of the peer support sessions as they wish.
4. Exit Interview: Participants will complete a follow-up semi-structured interview, held either in-person or virtually, conducted by the RA to ask about their experience receiving IPN support. Feedback will be elicited on what aspects of IPN support was helpful and what could be improved upon. Healthcare providers who work at clinic sites where recruitment took place will also be asked to take part in an individual interview about how the IPN service impacted their practice and care provision to Indigenous youth and their families.

ELIGIBILITY:
Inclusion Criteria:

* age 16-25 years;
* having chronic health condition of at least 3 months' duration that requires adult specialty follow-up care, including physical conditions (e.g., diabetes), mental health conditions (e.g., anxiety, depression), and/or developmental disorders (e.g., autism, fetal alcohol spectrum disorder);
* residing in Maskwacis or from the communities of Maskwacis but currently residing elsewhere;
* self-identified as an Indigenous person;
* reading level ≥ grade 6. For participants with developmental or intellectual delay (< grade 6 reading level), they may take part in the program alongside their caregiver(s).

Exclusion Criteria:

* not identifying as Indigenous
* not residing in Maskwacis

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Qualitative Analysis - Semi-structured interviews | 18 months
  Participants will complete a follow-up semi-structured interview, held either in-person or virtually, conducted by the RA to ask about their experience receiving IPN support. Feedback will be elicited on what aspects of IPN support was helpful and what could be improved upon. Healthcare providers who work at clinic sites where recruitment took place will also be asked to take part in an individual interview about how the IPN service impacted their practice and care provision to Indigenous youth and their families. All interviews will be recorded and transcribed verbatim, and NVivo software will be used for analysis. Thematic analysis will be used to extrapolate and systematically analyze patterns in the data generated by the qualitative data.

SECONDARY OUTCOMES:
Qualitative Analysis - Talking circles | 18 months
  Talking circles will be offered during the peer support sessions and facilitated by a community Elder. Participants will be asked about their transition experience moving from pediatric to adult care, how the IPN helped them (or didn't help them) to manage their health care and health condition, and how the IPN impacted their health and wellness. All interviews will be recorded and transcribed verbatim, and NVivo software will be used for analysis. Thematic analysis will be used to extrapolate and systematically analyze patterns in the data generated by the qualitative data.

CONTACTS AND LOCATIONS:
Locations (1):
- Stollery Children's Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No